CLINICAL TRIAL: NCT05707442
Title: Stent Implantation Versus Medical Therapy for Idiopathic IntracraniaL Hypertension (SIMPLE)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dapeng Mo, Clinical Professor of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2022042
Record Dates: First submitted 2022-12-25; First posted 2023-02-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Idiopathic Intracranial Hypotension; Venous Sinus Stenosis
Keywords: Idiopathic intracranial hypertension; Venous sinus stenosis; Stenting; Medical therapy; Randomized controlled trial
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent Implantation (Experimental): The endovascular procedure was performed under general anesthesia. Intravenous heparin was administered during the stent procedure to increase the activated clotting time to > 250 s. An 8F guiding catheter was delivered to the internal jugular vein near the skull base. A 6F Navien intermediate guide catheter was then placed into the distal transverse sinus near the torcula through the 8F guiding catheter. A microguidewire was navigated across the stenosis using a microcatheter, followed by the deployment of a self-expanding stent (eg, Precise or Wallstent) adjusted to the normal sinus venous diameter adjacent to the stenosis. Venography and manometry were performed after the procedure.
  Interventions: Procedure: Stent Implantation
- Medical Therapy (Active Comparator): The medical treatment consisted of acetazolamide (0.5-4 g/day) and short-term mannitol (bolus of 0.25-1 g/kg body weight) for a duration of about 1 week or repeated lumbar punctures to reduce intracranial pressure (20 mL each), as well as analgesics for headaches. The initial dosage of acetazolamide was 0.5 g daily in two divided doses, followed by dosage increases of one tablet every week up to a maximum dosage of 4 g/day. The dosage escalation was stopped if the participant had papilledema grade <1 in both eyes, unless the presence of other symptoms such as headache or tinnitus suggested that the dosage escalation should continue. The dosage for the participants who were unable to tolerate the study drug was decreased gradually to a minimum of one half tablet daily. In addition, the weight loss program included a low-calorie diet (≤425 kcal/day) with a target weight loss of approximately 5-10%.
  Interventions: Drug: Acetazolamide-based medical therapy; Behavioral: Weight loss

INTERVENTIONS:
Procedure: Stent Implantation — Aspirin (100 mg) and clopidogrel (75 mg) were administered 3-5 days before endovascular treatment. The endovascular procedure was performed under general anesthesia. Intravenous heparin was administered during the stent procedure to increase the activated clotting time to > 250 s. An 8F guiding catheter was delivered to the internal jugular vein near the skull base. A 6F Navien intermediate guide catheter was then placed into the distal transverse sinus near the torcula through the 8F guiding catheter. A microguidewire was navigated across the stenosis using a microcatheter, followed by the deployment of a self-expanding stent (eg, Precise or Wallstent) adjusted to the normal sinus venous diameter adjacent to the stenosis. Venography and manometry were performed after the procedure. Postoperatively, all patients received dual antiplatelet medications for 3 months and then received a single antiplatelet (either aspirin or clopidogrel).
  Arms: Stent Implantation
Drug: Acetazolamide-based medical therapy — The medical treatment consisted of acetazolamide (0.5-4 g/day) and short-term mannitol (bolus of 0.25-1 g/kg body weight) for a duration of about 1 week or repeated lumbar punctures to reduce intracranial pressure (20 mL each), as well as analgesics for headaches. The initial dosage of acetazolamide was 0.5 g daily in two divided doses, followed by dosage increases of one tablet every week up to a maximum dosage of 4 g/day. The dosage escalation was stopped if the participant had papilledema grade <1 in both eyes, unless the presence of other symptoms such as headache or tinnitus suggested that the dosage escalation should continue. The dosage for the participants who were unable to tolerate the study drug was decreased gradually to a minimum of one half tablet daily.
  Arms: Medical Therapy
Behavioral: Weight loss — The weight loss program included a low-calorie diet (≤425 kcal/day) with a target weight loss of approximately 5-10%.
  Arms: Medical Therapy

SUMMARY:
The aim of this study is to assess the efficacy of stent implantation versus medical therapy on idiopathic intracranial hypertension with venous sinus stenosis.

DETAILED DESCRIPTION:
The SIMPLE is a multicentered, prospective, randomized, open-label, blinded end-point clinical trial. A total of 74 patients with idiopathic intracranial hypertension (IIH) and venous sinus stenosis (VSS) for more than 2 months will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups (stenting or medical therapy) after offering informed content.

ELIGIBILITY:
Inclusion Criteria:

* Subject Eligibility Criteria

  1. Diagnosis of IIH by modified Dandy criteria about for more than 2 months
  2. Lumbar puncture opening pressure ≥250 mmH₂O within 6 weeks before enrollment
  3. Normal cerebrospinal fluid (CSF) composition
  4. Neuroimaging showing normal brain parenchyma without hydrocephalus, mass, or any structural lesion and no evidence of meningeal enhancement on CT or MRI
  5. Localized venous sinus stenosis (VSS) with stenotic degree ≥ 50% on DSA, and pressure gradient across stenosis ≥ 8 mmHg
  6. Patients or their relatives signed written informed consent
* Ophthalmic Eligibility Criteria:

  1. At least one eye had the presence of papilledema
  2. At least one eye of visual field loss: PMD ranging from - 2dB and below; decreased visual function on automated perimetry was reproducible with a false-positive rate of no more than 15%
  3. Visual acuity above 20 / 200 (≥ 39 letters)

Exclusion Criteria:

* Subject Exclusion Criteria

  1. Previous surgery for IIH, including optic nerve sheath fenestration (ONSF), CSF shunting, decompressive craniectomy or venous sinus stenting
  2. Progressive or rapid visual loss needed urgent surgical intervention; if delay>24-48 h consider interim lumbar drain (for rapid visual loss only).Surgical options to consider: CSF diversion or optic nerve sheath fenestration
  3. Visual loss due to other etiologies (eg, retinal drusen, retinal and optic neuropathy, cataracts, etc)
  4. Other condition requiring the use of diuretics, steroids or other drugs to reduce intracranial pressure
  5. DSA showed diffused venous sinus stenosis, cortical or deep vein stenosis
  6. A history of severe thyroid disease and iodine allergy
  7. Pregnant or lactating women
  8. Severe cardiopulmonary, liver or kidney failure
  9. Known hereditary or acquired haemorrhagic diathesis
  10. Known hereditary or acquired thrombophilia
  11. Platelet counts or coagulation abnormality
  12. Major surgery or severe trauma or any traumatic brain injury within the previous 14 days
  13. A history of cerebral hemorrhage, arteriovenous malformation, intracranial aneurysm or tumor
  14. Other life threatening illness (eg, advanced cancer) likely to lead to death within a few months; the physical, psychological and social status of patients may affect follow-up (eg, drug addiction, advanced malignant disease, no telephone, no family, etc); cannot tolerate general anesthesia
  15. Increased intracranial pressure due to other secondary factors
* Ophthalmic Exclusion Criteria:

  1. Current intraocular pressure > 28mmHg or previous intraocular pressure > 30mmHg
  2. Refractive error spherical power greater than -6.0D or +6.0D and astigmatism greater than 3.0D, except for the following cases:

     1. Myopia of - 6.0D to - 8.0D with the following: 1)There was no myopia related disease that can lead to decreased vision under the eyeground microscope (eg, scleral staphyloma, retinal thinning at the posterior pole, and moderate to severe disc tilt); 2) The patient wore contact lenses of appropriate degree for all visual field examinations.
     2. Hyperopia of +6.0D to +8.0D with the following: 1) The presence of a well characterized peri optic disc edematous halo, as opposed to crowded small optic discs or other features of decreased visual acuity associated with hyperopic changes, was at the discretion of the site investigator or reading center leader (or his designee); 2) The patient wore contact lenses of appropriate degree for all visual field examinations.
  3. Examination visible or past medical history known to have large optic disc drusen (persistent optic disc edema can present with small optic disc drusen, as low numbers are acceptable for inclusion and to be determined by the investigator to be unrelated to vision loss)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Perimetric Mean Deviation (PMD) | 6 months
  The change in perimetric mean deviation (PMD) from baseline to 6 month in the eye with the most severe visual loss at baseline.

SECONDARY OUTCOMES:
Cerebrospinal Fluid (CSF) Opening Pressure | 6 months
  The change in intracranial pressure measured by lumbar puncture opening pressure from baseline to 6 months.
Papilledema Grade: Frisén grade(0-5 scores,and higher scores mean worse outcome) | 6 months
  The change in papilledema measured by Frisén grade from baseline to 6 months
Retinal Nerve Fiber Layer Thickness | 6 months
  The change in thickness of retinal nerve fiber layer measured by optical coherence tomography (OCT) from baseline to 6 months.
Total Retinal Thickness | 6 months
  The change in thickness of total retina measured by optical coherence tomography (OCT) from baseline to 6 months.
Visual Acuity: National Eye Institute-Visual Function Questionnaire-25 (NEI-VFQ-25, minimum and maximum values: 0-100 points, higher scores mean a better visual function) | 6 months
  The change in vision measured by National Eye Institute-Visual Function Questionnaire-25 (NEI-VFQ-25) from baseline to 6 months.
Visual Acuity: 10-item neuro-ophthalmic supplement to the National Eye Institute-Visual Function Questionnaire-25 (NEI-VFQ-25) (minimum and maximum values: 0-100 points, higher scores mean a better visual function) | 6 months
  The change in vision measured by 10-item neuro-ophthalmic supplement to the National Eye Institute-Visual Function Questionnaire-25 (NEI-VFQ-25)from baseline to 6 months.
Headache: Headache Impact Test-6 (HIT-6, minimum and maximum values: 36-78 points, higher scores mean greater headache severity) | 6 months
  The change in headache measured by Headache Impact Test-6 (HIT-6) questionnaire from baseline to 6 months.
Pulsatile tinnitus: Tinnitus Handicap Inventory (THI, minimum and maximum values: 0-100 points, higher scores mean more serious tinnitus disability) | 6 months
  The change in pulsatile tinnitus from baseline to 6 months；pulsatile tinnitus was assessed using the Tinnitus Handicap Inventory (THI), which is a self-report measure that can be used in a busy clinical practice to quantify the impact of tinnitus on daily living.

OTHER OUTCOMES:
Functional health status and quality of life:EuroQol five dimensions questionnaire (EQ-5D,0-100,higher scores mean a better outcome) | 6 months
  The change in functional health status and quality of life measured by EuroQol five dimensions questionnaire (EQ-5D) from baseline to 6 months
Cost-effectiveness analysis (mean costs per patient) | 6 months
  The indicator of cost-effectiveness analysis refers to the mean costs per patient.
Cost-effectiveness analysis (quality-adjusted life years) | 6 months
  The indicator of cost-effectiveness analysis refers to the quality-adjusted life years.
Cost-effectiveness analysis (the cost saving per extra patient with a good outcome) | 6 months
  The indicator of cost-effectiveness analysis refers to the cost saving per extra patient with a good outcome.
Cost-effectiveness analysis (the cost saving per additional quality-adjusted life year) | 6 months
  The indicator of cost-effectiveness analysis refers to the cost saving per additional quality-adjusted life year.

CONTACTS AND LOCATIONS:
Overall Officials: Dapeng Mo, MD, Principal Investigator — Beijing Tiantan Hospital; Zhongrong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China